CLINICAL TRIAL: NCT03428945
Title: Hydroxychloroquine for Prevention of Abnormal Glucose Tolerance and Diabetes in Individuals At-risk for Type 1 Diabetes Mellitus (T1D)
Brief Title: Hydroxychloroquine in Individuals At-risk for Type 1 Diabetes Mellitus
Acronym: TN-22
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This trial has undergone a prespecified interim analysis which determined that this treatment provides no statistically significant delay in the onset of abnormal glucose tolerance or Type 1 Diabetes.
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Hydroxychloroquine; UC4DK117009 (NIH); UC4DK106993 (NIH)
Record Dates: First submitted 2018-01-24; First posted 2018-02-12 (Actual); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-07

CONDITIONS: Type1 Diabetes Mellitus
Keywords: TrialNet
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Treatment assignment (active drug: placebo) will be assigned in a parallel, randomized, 2:1 model. Assignment will be stratified based on prior treatment for T1D prevention and age.
Who Masked: Participant, Investigator
Masking Description: Active drug and placebo will be identical in appearance and packaging
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Experimental): Hydroxychloroquine compound for oral use
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Placebo tablet matching active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine for oral administration, dosed by weight
  Other Names: Plaquenil
  Arms: Hydroxychloroquine
Drug: Placebo — Placebo tablet identical to active drug
  Other Names: Inactive Drug
  Arms: Placebo

SUMMARY:
The study is a 2-arm, double blinded, multicenter, 2:1 randomized, placebo controlled clinical trial. Subjects will receive hydroxychloroquine or placebo and close monitoring for progression of T1D.

DETAILED DESCRIPTION:
This study is testing a medication, called hydroxychloroquine (HCQ) to assess safety and effectiveness to prevent individuals at risk of type 1 diabetes (T1D) from progressing to type 1 diabetes.

HCQ is approved by the U.S. Food and Drug Administration as a treatment for malaria, lupus, and rheumatoid arthritis. HCQ has been used extensively for treatment of autoimmune disease in adults, children, and during pregnancy. This medication has not previously been studied as a treatment to prevent T1D.

The goal of this study is to learn if HCQ can help prevent or delay progression from normal glucose tolerance (Stage 1) to abnormal glucose tolerance (Stage 2) or type 1 diabetes (Stage 3).

The study involves 5 visits in the first 6 months, then 1 visit every 6 months for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant in TrialNet Pathway to Prevention Study (TN01)
2. Age 3 years or greater at the time of randomization
3. Willing to provide informed consent
4. Normal glucose tolerance by OGTT within 7 weeks (no more than 52 days) of baseline
5. Two or more diabetes-related autoantibodies present on two separate samples
6. Weight of 12 kg or greater at screening
7. If a female participant with reproductive potential, willing to avoid pregnancy and undergo pregnancy testing prior to randomization and at each study visit
8. Anticipated ability to swallow study medication.

Exclusion Criteria:

1. Abnormal Glucose Tolerance or Diabetes
2. History of treatment with insulin or other diabetes therapies
3. Ongoing use of medications known to influence glucose tolerance
4. Ongoing or anticipated future use of medications known to have untoward interactions with hydroxychloroquine
5. Known hypersensitivity to 4-aminoquinoline compounds
6. G6PD deficiency
7. History of retinopathy
8. Have an active infection at time of randomization
9. Have serologic evidence of current or past HIV, Hepatitis B (positive for Hepatitis B core antibody or surface antigen), or Hepatitis C infection
10. Deemed unlikely or unable to comply with the protocol or have any complicating medical issues, including prolonged QT interval, a disease previously or likely in the future to require immunosuppression, or abnormal clinical laboratory results that interfere with study conduct or cause increased risk.
11. Deemed unlikely or unable to comply with the protocol or have any complicating medical issues, including prolonged QT interval, a disease previously or likely in the future to require immunosuppression, or abnormal clinical laboratory results that interfere with study conduct or cause increased risk.
12. Be pregnant or breastfeeding.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Greenbaum, MD, Study Chair — Type 1 Diabetes TrialNet
Locations (51):
- United States (37):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Barbara Davis Center, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - USF Diabetes Center, Tampa, Florida
  - Emory Children's Center, Atlanta, Georgia
  - St. Luke's Humphreys Diabetes Center, Boise, Idaho
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - University of Chicago, Chicago, Illinois
  - Indiana University - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky/UK Healthcare, Lexington, Kentucky
  - University of Louisville Pediatric Endocrinology, Louisville, Kentucky
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Palm Research Center, Inc., Las Vegas, Nevada
  - UBMD Pediatrics, Buffalo, New York
  - Columbia University, New York, New York
  - Joslin Center at SUNY Upstate Medical University, Syracuse, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The University of Oklahoma, Oklahoma City, Oklahoma
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Endocrinology Specialist / Greenville Health System, Greenville, South Carolina
  - GHS - Pediatric Endocrinology, Greenville, South Carolina
  - Sanford Children's Specialty Clinic, Sioux Falls, South Dakota
  - Vanderbilt Eskind Diabetes Clinic, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Benaroya Research Institute, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Women's and Children's Hospital, Adelaide, North Adelaide, South Australia
  - Walter and Eliza Hall Institute of Medical Research, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (3):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital For Sick Kids, Toronto, Ontario
  - IWK Health Center, Halifax
- San Raffaele Hospital, Milan, Italy
- Skane University Hospital, Malmo, Sweden
- United Kingdom (5):
  - Royal Devon and Exeter Hospital, Exeter, Devon
  - Plymouth Diabetes Clinical Research Unit, Plymouth, Devon
  - Harrogate and District NHS Foundation Trust, Harrogate, North Yorkshire
  - University of Bristol, Bristol, UK
  - Nottingham University Hospitals, Nottingham

REFERENCES:
- See also: TrialNet Public Website — http://www.trialnet.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydroxychloroquine | Placebo
Started | 183 | 90
Completed | 168 | 77
Not Completed | 15 | 13
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Placebo | Total
Number analyzed (Participants) | 183 | 90 | 273
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 165 | 77 | 242
  Between 18 and 65 years | 18 | 13 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 11.7 [8.3 to 15.6] | 10.9 [8.2 to 15.7] | 11.3 [8.3 to 15.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 33 | 94
  Male | 122 | 57 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 4 | 19
  Not Hispanic or Latino | 162 | 82 | 244
  Unknown or Not Reported | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 171 | 83 | 254
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 7 | 16
  Sweden | 1 | 0 | 1
  United States | 155 | 72 | 227
  United Kingdom | 2 | 2 | 4
  Italy | 0 | 2 | 2
  Australia | 13 | 7 | 20
  Finland | 3 | 0 | 3
Relationship to person with Type 1 Diabetes [Count of Participants; unit: Participants]
  More than one first degree relative | 15 | 6 | 21
  Sibling(s) | 100 | 48 | 148
  Offspring | 6 | 5 | 11
  Parent(s) | 42 | 22 | 64
  Second Degree Relative | 9 | 6 | 15
  Third Degree Relative | 1 | 0 | 1
  No Relatives | 10 | 3 | 13
Autoantibodies positive [Count of Participants; unit: Participants]
  1 positive Autoantibody | 2 | 1 | 3
  2 positive Autoantibodies | 35 | 23 | 58
  3 positive Autoantibodies | 39 | 24 | 63
  4 positive Autoantibodies | 46 | 18 | 64
  5 positive Autoantibodies | 61 | 24 | 85

OUTCOME MEASURES:

1. Primary Outcome: Change From Treatment Assignment Glucose Tolerance to Abnormal Glucose Tolerance or Diabetes
Description: The primary outcome is the time in months from random treatment assignment to the development of confirmed abnormal glucose tolerance or clinical diabetes.
Time Frame: Glucose tolerance is measured every 6 months for up to 4 years
Population: Participants included in the time-to-event analysis
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 168 | 83
Months | 19.7 [10.6 to 36.2] | 18.8 [9.9 to 33.1]

ADVERSE EVENTS:
Time Frame: Duration of study from screening to last visit encompassing each participant's duration of time in the study no more than 4 years with an average duration prior to study termination of 23.9 months.
Description: Adverse Events were defined using the Common Terminology Criteria for Adverse Events (CTCAE)
Arm/Group | Hydroxychloroquine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/90
Serious Adverse Events (participants affected / at risk) | 5/183 | 1/90
Other Adverse Events (participants affected / at risk) | 125/183 | 61/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=183) | Placebo (N=90)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 1 (1) — Bruising
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=183) | Placebo (N=90)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 2 (6) | 1 (1)
Vision decreased (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (3) | 4 (5)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6) | 0 (0)
Fever (General disorders) | 5 (7) | 0 (0)
Flu like symptoms (General disorders) | 2 (2) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (3) | 4 (5)
Pain (General disorders) | 2 (2) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (2) | 2 (2)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 2 (2) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Esophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 3 (4) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 29 (33) | 13 (14)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 4 (4) | 5 (5)
Penile infection (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 3 (3) | 4 (4)
Sinusitis (Infections and infestations) | 11 (13) | 5 (5)
Skin infection (Infections and infestations) | 3 (3) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 16 (21) | 7 (10)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 8 (8) | 3 (3)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 8 (19) | 5 (5)
Venous injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (3) | 3 (6)
Creatinine increased (Investigations) | 4 (4) | 0 (0)
Investigations - Other, specify (Investigations) | 6 (6) | 3 (3)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 32 (56) | 26 (41)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 3 (3) | 1 (1)
White blood cell decreased (Investigations) | 4 (4) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 6 (8) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (7) | 3 (4)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 4 (6) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 4 (5) | 3 (4)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (6)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 16 (19) | 5 (7)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 10 (12) | 3 (4)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Interim analysis completed prompted the DSMB's decision to terminate the protocol early limiting the originally planned follow up period for participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT03428945/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT03428945/SAP_001.pdf